CLINICAL TRIAL: NCT01238627
Title: Bioequivalence Between Two Oral Nicotine Sublingual Tablets, 2 mg and 4 mg - A Study in Healthy Smokers
Brief Title: Bioequivalence Between Two Oral Nicotine Sublingual Tablets, 2 mg and 4 mg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NICTDP1064-A6431115; 2007-002180-27 (EudraCT Number)
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nicotine Sublingual Tablet Mint (NSTM)-2 (Experimental): Experimental 2 mg NSTM
  Interventions: Drug: Nicotine Sublingual Tablet Mint (NSTM)
- Microtab-2 (Active Comparator): 2 mg Nicotine tablet
  Interventions: Drug: Marketed Nicotine Tablet
- NSTM-4 (Experimental): Experimental 4 mg Nicotine Sublingual Tablet Mint
  Interventions: Drug: Nicotine Sublingual Tablet Mint (NSTM)
- Microtab-4 (Active Comparator): 2 x 2 mg Nicotine tablet
  Interventions: Drug: Marketed Nicotine Tablet

INTERVENTIONS:
Drug: Nicotine Sublingual Tablet Mint (NSTM) — A single dose of an experimental NSTM, with a 36-hour washout between visits
  Other Names: Not marketed
  Arms: NSTM-4; Nicotine Sublingual Tablet Mint (NSTM)-2
Drug: Marketed Nicotine Tablet — A single dose of a marketed Nicotine Replacement Therapy (NRT), with a 36-hour washout between visits
  Other Names: Nicorette® Microtab
  Arms: Microtab-2; Microtab-4

SUMMARY:
The purpose of this study is to assess the bioequivalence between two oral nicotine sublingual tablets, 2 mg and 4 mg.

DETAILED DESCRIPTION:
The study is a single-dose, randomized, 2 x two-way cross-over study. The investigational products will be given as single doses at separate visits. Periods without Nicotine Replacement Therapy (NRT), lasting for at least 36 hours, will separate treatment visits. Blood will be sampled at each treatment visit for pharmacokinetic analyses pre-dose, and at 5, 10, 15, 20, 30, and 45 minutes, as well as 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 10 hours after start of product administration. The time until complete product dissolution will be recorded. Subjects will also be monitored to capture any adverse events that may occur. The trial is open in the sense that subjects and study personnel will be aware of what product is administered at a given visit. However, the treatment labels will not be known by the people performing bioanalysis or analyzing pharmacokinetic data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, smoking at least 10 cigarettes daily during at least one year preceding inclusion and Body Mass Index (BMI) between 17.5 and 30.0 kg/m2.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 months preceding the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | During 10 hours post-dose
  Cmax, which is the maximum observed plasma concentration after a dose is administered, measured in nanograms/milliliter (ng/mL)
Area Under the Curve (AUC)(0-t) | During 10 hours post-dose
  Bioavailability within the Set Period [AUC(0-t)] is the area under the plasma concentration verses time curve from start of drug administration until the time of the last measurable plasma concentration, calculated as hour * nanograms (ng) per milliliter (mL).
AUC(0-∞) | 10 hours post-dose
  AUC (0-∞) is the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time. It is obtained from calculating AUC (0-t) plus AUC (t-∞).

SECONDARY OUTCOMES:
Product Dissolution Time | During 10 hours post-dose
  Product Dissolution Time is the time from administration until the investigational products were completely dissolved.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- McNeil AB Clinical Pharmacology R&D, Lund, Sweden